CLINICAL TRIAL: NCT02989376
Title: Emergent Carotid Ultrasound in Hyperacute Cerebral Vessel Occlusion for Selecting Patients to be Treated With Endovascular Clot Retrieval Treatment
Brief Title: Carotid Duplex Ultrasound for Selecting Patients for Endovascular Thrombectomy in Acute Stroke Patients
Acronym: ECHO-SELECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryo Itabashi (Other)
Responsible Party: Sponsor-Investigator, Ryo Itabashi, Department chair of Stroke Neurology, Kohnan Hospital
Organization: Kohnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KohnanSN01
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

ARMS (1):
- carotid duplex ultrasound (Experimental): Single arm study. After detection of occluded vessels by vascular imaging using carotid duplex ultrasound, digital subtraction angiography is immediately performed before acute endovascular treatment.
  Interventions: Procedure: After detection of occluded vessels by vascular imaging using carotid duplex ultrasound, digital subtraction angiography is immediately performed before acute endovascular treatment.

INTERVENTIONS:
Procedure: After detection of occluded vessels by vascular imaging using carotid duplex ultrasound, digital subtraction angiography is immediately performed before acute endovascular treatment. — When the ratio of the end diastolic velocity in the common carotid arteries is greater than 1.4 or the diastolic flow in the internal carotid artery is not detected by vascular imaging using carotid duplex ultrasound, digital subtraction angiography is immediately performed before acute endovascular treatment. If vessel occlusion is not detected by carotid duplex ultrasound, additional vascular imaging including MR angiography or CT angiography is considered.

SUMMARY:
The aim of this study is to address the usefulness of carotid duplex ultrasound as vascular imaging for selecting acute stroke patients for endovascular thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Endovascular treatment can be initiated within 6 hours of symptom onset.
* ASPECTS of >=6 is diagnosed by two or more stroke physicians.
* The end diastolic velocity in the common carotid arteries or internal carotid artery is evaluated by carotid duplex ultrasound
* NIHSS score of >=6.
* Age>=18 years.
* Written informed consent is obtained.

Exclusion Criteria:

* Pre-stroke modified Rankin Scale (mRS) score >=2.
* Difficulties to evaluate ASPECTS on initial CT.
* Difficulties to groin puncture.
* History of severe allergic reaction to contrast medium.
* End stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | at 90 days after onset

CONTACTS AND LOCATIONS:
Overall Officials: Ryo Itabashi, MD, Principal Investigator — Kohnan Hospital
Locations (1):
- Kohnan hospital, Sendai, Miyagi, Japan